CLINICAL TRIAL: NCT00167401
Title: A Phase II Trial of One-Cycle Induction Chemotherapy Followed by Pulsed Docetaxel and Concurrent Radiation for Non-Small Cell Lung Cancer
Brief Title: Trial of Chemotherapy Followed by Pulsed Docetaxel and Concurrent Radiation for Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Yuhchyau Chen, MD, Ph.D, University of Rochester, Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: URCC 1500; Aventis 12083-Chen
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2009-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: docetaxel
Drug: cisplatin
Procedure: radiation treatment

SUMMARY:
The University of Rochester Cancer Center (URCC) is conducting a research study at Highland Hospital and Strong Memorial of lung cancer patients whose tumors cannot be surgically removed. The usual treatment for this stage of cancer is chemotherapy (treatment with drugs) combined with radiation (chemo-radiation). Because of the risk of spread to other organs, patients with your stage of disease are also often treated with additional chemotherapy, either before or after the chemo-radiation treatment. The best timing and number of treatments for this additional chemotherapy has not been clearly established. The purpose of this study is to help determine if a single treatment with two chemotherapy drugs, followed by radiation and low-dose chemotherapy is an effective way to treat patients with lung cancer. The side effects of this treatment and your quality of life while on the study will also be studied. Eighteen will participate in this study locally.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed non-small cell lung cancer.

Clinical or pathologic stage IIIA (T1-3N2M0, T3N1M0) and IIIB (Any T N3M0, T4 Any N M0) diseases according to the American Joint Committee of Cancer criteria (Appendix I). Patients with malignant pleural effusion will be excluded.

The primary tumor must be radiographically measurable with bi-dimensionally measurable disease

Age > 18.

Karnofsky performance status > 70 (Appendix II).

FEV1 sufficient for patients to tolerate radiation therapy, which is at the discretion of the radiation oncologist, usually > 800 ml, but may be higher or lower depending on the volume of radiotherapy portal, which is a variable of the tumor extent.

WBC > 3000; platelet count > 100,000; absolute neutrophil counts > 1,000; hemoglobin ≥ 8.0 g/dl; serum creatinine < 1.5 mg/dl or creatinine clearance >60 ml/min. Laboratory values must be obtained < 3 weeks prior to registration.

Patients with equivocal enlargement of adrenal gland(s) on CT scan, or a few equivocal regional or distant lesions on any imaging studies need further imaging study or biopsy to rule out distant metastasis.

Transaminases (SGOT and/or SGPT) may be up to 2.5 x institutional upper limit of normal (ULN) if alkaline phosphatase is < ULN, or alkaline phosphatase may be up to 4 x ULN if transaminases are < ULN. However, patients who have both transaminase elevation > 1.5 x ULN and alkaline phosphatase > 2.5 x ULN are not eligible for this study (due to decreased clearance of docetaxel and increased risk of toxicity).

Pre-existing neuropathy must be grade I or less.

A signed informed consent.

Women of childbearing potential must have a negative pregnancy test.

Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for a reasonable period thereafter.

Exclusion Criteria:

Patients with distant metastasis (stage IV disease).

Patients without measurable disease.

Patients with medical contraindication to chemotherapy or radiotherapy.

Patients with myocardial infarction within the preceding six months or symptomatic heart disease, including angina, congestive heart failure, uncontrolled arrhythmia.

Patients with bilirubin elevated above institutional upper limit of normal (ULN) must be excluded.

Women who are pregnant or breast feeding are not eligible.

Patients with a history of severe hypersensitivity reaction to Taxotere® or other drugs formulated with polysorbate 80 must be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-02; Primary Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuhchyau Chen, MD, Ph.D, Principal Investigator — Universtiy of Rochester, Dept of Radiation Oncology
Locations (1):
- University of Rochester, Dept. Radiation Oncology, Rochester, New York, United States